CLINICAL TRIAL: NCT01345630
Title: A Multicenter, Randomized, Double-Blind, Comparative Trial Of Maraviroc + Darunavir/Ritonavir Versus Emtricitabine/Tenofovir + Darunavir/Ritonavir For The Treatment Of Antiretroviral-Naive Hiv-Infected Patients With Ccr5-Tropic Hiv-1
Brief Title: Comparative Trial Of Maraviroc Versus Emtricitabine/Tenofovir Both With Darunavir/Ritonavir In Antiretroviral-Naive Patients Infected With CCR5 Tropic HIV 1
Acronym: MODERN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4001095; 2010-021785-30 (EudraCT Number)
Record Dates: First submitted 2011-04-27; First posted 2011-05-02 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: HIV-1
Keywords: Double-blind; comparative; trial; maraviroc; versus; emtricitabine/tenofovir; both with darunavir/ritonavir; antiretroviral-naive; Ccr5 tropic; Hiv 1; patients.
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Darunavir; Ritonavir; Emtricitabine; Tenofovir

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc (Experimental): Maraviroc 150 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for emtricitabine/tenofovir once daily.
  Interventions: Drug: Maraviroc; Drug: darunavir/ritonavir 800/100 mg; Drug: placebo for maraviroc
- Emtricitabine/tenofovir (Active Comparator): Emtricitabine/tenofovir 200/300 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for maraviroc once daily.
  Interventions: Drug: Emtricitabine/tenofovir; Drug: placebo for emtricitabine/tenofovir

INTERVENTIONS:
Drug: Maraviroc — Maraviroc tablet 150 mg once daily for 96 weeks.
  Other Names: Selzentry, Celsentri
  Arms: Maraviroc
Drug: Emtricitabine/tenofovir — Emtricitabine/tenofovir tablet 200/300 mg once daily for 96 weeks.
  Other Names: Truvada
  Arms: Emtricitabine/tenofovir
Drug: darunavir/ritonavir 800/100 mg — darunavir/ritonavir 800/100 mg
  Arms: Maraviroc
Drug: placebo for emtricitabine/tenofovir — placebo for emtricitabine/tenofovir
  Other Names: Truvada
  Arms: Emtricitabine/tenofovir
Drug: placebo for maraviroc — placebo for maraviroc
  Other Names: Selzentry, Celsentri
  Arms: Maraviroc

SUMMARY:
The purpose of this study is to assess whether maraviroc administered once daily is non-inferior to emtricitabine/tenofovir also administered once daily each in combination with darunavir/ritonavir in the treatment of antiretroviral-naive patients as evaluated at Week 48 of treatment.

DETAILED DESCRIPTION:
The study was terminated on October 8, 2013 following a preliminary review of the Week 48 primary efficacy data by the study's external independent Data Monitoring Committee (DMC). The DMC assessed the data as demonstrating significant differences between the treatment arms in virologic responses and failures. The DMC recommended and the Sponsor concurred that the study be terminated because of the inferior efficacy of the Maraviroc arm as compared to the comparator arm (Emtricitabine/Tenofovir).

ELIGIBILITY:
Inclusion Criteria:

* Plasma HIV-1 RNA equal to or greater than 1,000 copies/mL measured at the Screening Visit.
* CD4 count equal to or greater than 100 cells/mm3 at Screening.
* Have only R5 HIV 1 at Screening as verified by a randomized tropism assay.

Exclusion Criteria:

* Prior treatment with any other HIV antiretroviral therapy for more than 14 days at any time.
* Any evidence of genotypic/phenotypic resistance to darunavir, tenofovir, and emtricitabine.
* CXCR4 using virus detected using randomized tropism determination or repeated failure to obtain an interpretable tropism result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (175):
- United States (82):
  - University of Alabama at Birmingham - 1917 Research Clinic, Birmingham, Alabama
  - Health Services Center, Hobson City, Alabama
  - Kaiser Permanente, Hayward, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Dr. Anthony Mills, MD, Inc., Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - University of California Davis Research, Sacramento, California
  - TICON I Research Clinic (DEXA Scan only), Sacramento, California
  - Kaiser Hospital Sacramento, Sacramento, California
  - Synarc Inc., San Francisco, California
  - Investigational Drugs Pharmacy, San Francisco, California
  - Kaiser Permanente - Clinical Trials Unit, San Francisco, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Kaiser Permanente, Union City, California
  - University of Colorado Denver - University of Colorado Hospital, Aurora, Colorado
  - Kaiser Permanente of Colorado, Denver, Colorado
  - Yale - New Haven Hospital Nathan Smith Clinic, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Circle CARE Center, Norwalk, Connecticut
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Broward Health - Comprehensive Care Center, Fort Lauderdale, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - The Kinder Medical Group, Miami, Florida
  - UMHC/Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami AIDS Clinical Research Unit, Miami, Florida
  - University of Miami, Miami, Florida
  - Community AIDS Resource Inc dba Care Resource, Miami, Florida
  - Miami Research Associates, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Infectious Diseases Associates of Northwest Florida, PA, Pensacola, Florida
  - St. Joseph's Hospital Diagnostic Center, Tampa, Florida
  - University of South Florida Health-HIV Clinical Research Unit, Tampa, Florida
  - Infectious Disease Research Institute, Inc., Tampa, Florida
  - Osteoporosis Care Center, Tampa, Florida
  - Quest Diagnostic Laboratory, Tampa, Florida
  - Rowan Tree Medical, PA, Wilton Manors, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - DeKalb Medical Diagnostic Breast Center, Decatur, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Northwestern University/NMH, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - University of Iowa, University of Hospitals and Clinics - Division of Infectious Disease, Iowa City, Iowa
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Be Well Medical Center, PC, Berkley, Michigan
  - University Physicians Group, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University College of Osteopathic Medicine - Department of Internal Medicine, East Lansing, Michigan
  - Biomedical and Health Institutional Review Board, East Lansing, Michigan
  - Ingham County Health Department, Lansing, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Kansas City Free Health Clinic, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Brandywine Common, Neptune City, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Beth Israel Medical Center - AIDS Clinical Trials Unit, New York, New York
  - AIDS Community Research Initiative of America (ACRIA), New York, New York
  - Research Across America, New York, New York
  - Dr. Howard A. Grossman, M.D., New York, New York
  - AIDS Care, Rochester, New York
  - New York Medical College, Valhalla, New York
  - I.D. Consultants, P.A., Charlotte, North Carolina
  - (DEXA Scan Facility) East Carolina University Brody Outpatient Center, Greenville, North Carolina
  - East Carolina University Division of Infectious Diseases, Greenville, North Carolina
  - University of Cincinnati - Department of Internal Medicine, Cincinnati, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - Central Texas Clinical Research, Austin, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, PA, Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - The Office of Dr. Gordon E. Crofoot, M.D., PA, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
- Australia (7):
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Holdsworth House General Practice, Darlinghurst, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Surry Hills, New South Wales
  - Brisbane Sexual Health and HIV Service, Brisbane, Queensland
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Clinical Research Unit, Infectious Diseases, Melbourne, Victoria
- AKH Wien Universitaetsklinik fuer Dermatologie, Vienna, Austria
- Belgium (6):
  - Instituut voor Tropische Geneeskunde, Antwerp
  - C.H.U. St-Pierre, Brussels
  - Hôpital Universitaire Erasme, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - C.H.U. Sart-Tilman, Liège
- Canada (7):
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - The Ottawa Hospital-Riverside Campus, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Maple Leaf Research / Maple Leaf Medical Clinic, Toronto, Ontario
  - University Health Network / Toronto General Hospital, Toronto, Ontario
  - Clinique Medicale L'Actuel, Montreal, Quebec
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
- Denmark (3):
  - Hvidovre Hospital, Infektionsmedicinsk afd., Hvidovre
  - Rigshospitalet, Epidemiklinikken, Koebenhavn OE
  - Odense Universitetshospital, Odense
- Infektiosairauksien poliklinikka,HUS Auroran sairaala, rakennus 5, 1. krs, Helsinki, Finland
- France (14):
  - CHR d'Orleans la Source, Orléans, Cedex 02
  - Hopital Saint Antoine, Paris, Cedex 12
  - Hopital Bichat, Paris, Cedex 18
  - Hopital Saint-andre, Bordeaux, France
  - Hopital Henri Mondor, Créteil
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Hopital de la Croix Rousse, Lyon
  - Hopital Gui de Chauliac, Montpellier
  - CHU de Nantes - Hotel Dieu, Nantes
  - Hôpital de la Pitié Salpétrière, Paris
  - Hopital Tenon, Service des Maladies Infectieuses, Paris
  - Hopital Saint-Louis, Paris
  - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (12):
  - Praxis Christiane Cordes, Berlin
  - Studiengesellschaft mbH Gubener 37, Berlin
  - EPIMED - Gesellschaft fuer epidemiologische und klinische Forschung in der Medizin mbH, Berlin
  - Universitaetsklinikum Bonn, Immunologische Ambulanz HIV, Bonn
  - Klinikum der Universitaet zu Koeln, Klinik I fuer Innere Medizin, Cologne
  - Klinikum der J.W. Goethe-Universitaet, Medizinische Klinik II, Frankfurt am Main
  - InfektioResearch GmbH & Co. KG, Frankfurt am Main
  - ifi - Studien und Projekte GmbH, Hamburg
  - ICH - Study - Center GmbH & Co. KG, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - MUC Research Group GbR, München
  - Ludwig-Maximilians-Universitaet, Medizinische Poliklinik - Klinikum Innenstadt, München
- Egyesitett Szent Istvan és Szent Laszlo Korhaz-Rendelointezet, Budapest, Hungary
- Ospedale San Raffaele, Milan, Italy
- University Medical Center Utrecht, Utrecht, Netherlands
- Poland (3):
  - Wojewodzki Szpital Obserwacyjno - Zakazny im. Tadeusza Browicza, Bydgoszcz
  - SPZOZ Wojewodzki Szpital Zakazny, Warsaw
  - EMC Instytut Medyczny S.A. Przychodnia przy ul. Lowieckiej, Wroclaw
- Portugal (4):
  - Hospital Prof. Doutor Fernando Fonseca E.P.E., Amadora, Portugal
  - Centro Hospitalar de Lisboa - Zona Central - Hospital Santo António Capuchos, Lisbon
  - Hospital Sta. Maria, Lisbon
  - Hospital São João, Porto
- Puerto Rico (6):
  - Innovative Care PSC, Bayamón, PR
  - Ararat Research Center, Ponce, PR
  - Medical Center University Hospital, Rio Piedras, PR
  - Clinical Research Puerto Rico, San Juan, PR
  - HOPE Clinical Research, San Juan, PR
  - University of Puerto Rico Medical Sciences Campus, Rio Piedras
- Spain (9):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia - Hospital Provincial, Córdoba, Cordoba
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario de La Paz, Madrid, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville, Sevilla
- Sweden (4):
  - SU Ostra sjukhuset, Infektionsmottagningen, Gothenburg
  - Skanes Universitetssjukhus, Malmo
  - Sodersjukhuset, Venhalsan, Stockholm
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- Switzerland (4):
  - Universitaetsspital Basel Infektiologie und Spitalhygiene, Basel
  - Inselspital Universitaetsklinik fuer Infektiologie, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitatsspital Zurich, Zurich
- United Kingdom (9):
  - Dept of Sexual Health & HIV Medicine, Birmingham
  - HIV Research Department, Elton John Centre, Brighton
  - Regional Infectious Diseases Unit, Edinburgh
  - Grahame Hayton Unit, Ambrose King Centre, Royal London Hospital,, London
  - Ian Charleson Day Centre, Royal Free Hospital, London
  - Queen Elizabeth Hospital, London
  - St Stephen's Centre, Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Centre for Sexual Health & HIV Research, University College London, London
  - Department of Infectious Diseases & Tropical Medicine, Pennine Acute Trust Hospitals, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001095&StudyName=Comparative%20Trial%20Of%20Maraviroc%20Versus%20Emtricitabine/Tenofovir%20Both%20With%20Darunavir/Ritonavir%20In%20Antiretroviral-Naive%20Patients%20Infected%20With%20Ccr5%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 1423 participants were screened and 813 participants randomized in the study. A total of 797 participants were treated (396 were treated in the maraviroc + darunavir/ritonavir [MVC+DRV/r] group and 401 in the emtricitabine/tenofovir + darunavir/ritonavir [FTC/TDF+DRV/r] group). The study was conducted in 138 sites in 18 countries.
Pre-assignment Details: Participants were randomized to undergo either genotype testing or enhanced Trofile assay (ESTA) in a 1:1 ratio. Among participants who were identified as being infected with R5 tropic HIV-1 by either testing methods, 813 were randomized in a 1:1 ratio to receive 96-week treatment either in the MVC+DRV/r arm or in the FTC/TDF+DRV/r arm.
Groups:
- MVC+DRV/r: Participants infected with R5 HIV-1 received oral tablets of Maraviroc 150 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for emtricitabine/tenofovir once daily.
- FTC/TDF+DRV/r: Participants infected with R5 HIV-1 received oral tablets of emtricitabine/tenofovir 200/300 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for maraviroc once daily.
Period: Overall Study
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Started | 396 | 401
Completed | 35 | 42
Not Completed | 361 | 359
Not completed — Adverse Event | 22 | 23
Not completed — Lost to Follow-up | 17 | 16
Not completed — Protocol Violation | 4 | 1
Not completed — Medication error without associated AE | 0 | 1
Not completed — Study terminated by sponsor | 254 | 285
Not completed — Other reasons | 6 | 8
Not completed — Withdrawn due to pregnancy | 1 | 2
Not completed — No longer willing to participate | 9 | 12
Not completed — Insufficient clinical response | 48 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r | Total
Number analyzed (Participants) | 396 | 401 | 797
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (10.9) | 36.2 (10.9) | 37.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 360 | 367 | 727

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/mL.
Description: The proportion of participants who achieved HIV-1 RNA <50 copies/mL at week 48 was assessed according to Food and Drug Administration's (FDA's) Missing, Switch, Discontinuation'=Failure (MSDF) Snapshot algorithm. The algorithm used the plasma HIV-1 RNA in the Week 48 visit window, followed the "virology-first principle" and considers a participant who has a missing plasma HIV-1 RNA, or switches to prohibited ARV regimen or discontinues from the study or study drug for any reason, or dies, as a failure.
Time Frame: Week 48
Population: The Full Analysis Set (FAS) consisted of all randomized participants who received at least one dose of the study drug. The missing value was imputed per FDA's MSDF Snapshot algorithm as described under "Outcome Measure Description" above.
Measure: Number; unit: Percentage of participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
Percentage of participants | 77.3 | 86.8
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; The difference in the percentages between the maraviroc and the emtricitabine/tenofovir treatment arms and the 2-sided 95% confidence interval for the difference was provided using the stratum-adjusted Mantel-Haenszel (MH) method over the two assays and the screening plasma HIV-1 RNA levels (>=100,000 copies/mL or <100,000 copies/mL). The sample size was chosen to yield a power of ≥90%. The 95% CIs and mean difference (final values) are presented as percentages above; Test type: Non-Inferiority or Equivalence — For the analysis of the primary endpoint conducted at Week 48, the alternative hypothesis was to test for non-inferiority of MVC+DRV/r to FTC/TDF+DRV/r with a non-inferiority margin of -10%; Mean Difference (Final Values) = -9.54, 95% CI 2-sided [-14.83 to -4.24]

2. Secondary Outcome: Frequency of Adverse Events (AE).
Description: Number of participants with treatment-emergent non serious AEs
Time Frame: Week 96
Population: Safety Analysis Set was the same as the FAS consisting of all randomized participants who received at least one dose of the study drug but analyzed as realized for tropism assay and treatment.
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
participants | 360 | 365

3. Secondary Outcome: Number of Participants With Grade 3 or 4 AEs
Description: Number of participants with grade 3 or 4 AEs are presented here.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
participants | 65 | 71

4. Secondary Outcome: Number of Participants Who Discontinued Due to AEs
Description: Number of participants who discontinued due to AEs are reported here. Three participants (two from the MVC+DRV/r arm and one from the FTC/TDF+DRV/r arm) were not considered as discontinued due to AE because other reasons for discontinuation were prioritized for these participants.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
participants | 22 | 23

5. Secondary Outcome: Number of Treatment-related AEs
Description: Number of treatment-related AEs are presented here.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: events
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
events | 316 | 361

6. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events
Description: Total number of participants with treatment-emergent serious adverse events are reported
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
participants | 41 | 40

7. Secondary Outcome: Number of Participants With Abnormal Laboratory Values
Description: Number of participants with laboratory abnormalities are reported
Time Frame: Week 96
Population: Safety Analysis Set was the same as the FAS consisting of all randomized participants who received at least one dose of the study drug but analyzed as realized for tropism assay and treatment. One participant was not analyzed for laboratory data as the collection date for all lab data was less than the first active therapy date.
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 400
participants
  Normal Baseline | 210 | 205
  Abnormal Baseline | 111 | 101

8. Secondary Outcome: Severity of Abnormal Laboratory Values
Description: Number of participants who had clinically significant laboratory abnormalities of Grade 3 and Grade 4 according to DAIDS. Abnormality incidence of highest grade was reported for a labcode for each individual participant.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
participants
  Alanine Aminotransferase (ALT) (n=396, 400) | 9 | 6
  Alkaline Phosphatase (n=396, 400) | 1 | 0
  Amylase (n=396, 400) | 5 | 13
  Aspartate Aminotransferase (AST) (n=396, 400) | 11 | 7
  Blood Urea Nitrogen (BUN) (n=396, 400) | 3 | 5
  Calcium (n=396, 400) | 7 | 10
  Creatine Kinase (n=396, 400) | 18 | 22
  Hemoglobin (n=396, 400) | 4 | 2
  LDL Cholesterol (n=396, 400) | 50 | 24
  Lipase (n=116, 122) | 3 | 10
  Lymphocytes (Abs) (n=396, 400) | 2 | 2
  Phosphate (n=396, 400) | 5 | 12
  Platelets (n=396, 400) | 5 | 1
  Potassium (n=396, 400) | 3 | 2
  Sodium (n=396, 400) | 2 | 0
  Total Bilirubin (n=396, 400) | 3 | 1
  Total Neutrophils (Abs) (n=396, 400) | 6 | 2
  Triglycerides (n=396, 400) | 4 | 6
  Uric Acid (n=396, 400) | 0 | 2
  White Blood Cell Count (n=396, 400) | 1 | 0
  Creatinine (n=396, 400) | 0 | 1

9. Secondary Outcome: The Relationship Between the Proportion of Participants With Plasma HIV-1 RNA <50 Copies/mL at the Week 48 and the Screening Tropism Test (Genotype Test or ESTA).
Description: The relationship of the proportion of participants achieving HIV-1 RNA <50 copies/mL at Week 48 with the screening tropism test for the MVC containing regimen was analyzed. Virologic response for a participant at Week 48 was derived using the FDA's Snapshot MSDF algorithm. Difference in proportions of patients with plasma HIV-1 RNA <50 copies/mL at week 48 between the maraviroc and the emtricitabine/tenofovir treatment arms, with two-sided 95% confidence interval, among patients who are R5 by genotype (including some who were originally randomized to ESTA and are R5 by genotype upon retesting), were calculated via the Maximum Likelihood method. The estimate was adjusted for the screening plasma HIV RNA level (<100,000 vs. ≥100,000) copies/mL via the Mantel Haenszel (MH) method.
Time Frame: Week 48
Population: The FAS consisted of all randomized participants who received at least one dose of the study drug.
Measure: Number; unit: proportion of participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
proportion of participants | 0.8047 (0.0238) | 0.8797 (0.0187)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; The difference in proportions of patients with plasma HIV-1 RNA <50 copies/mL at Week 48 between the [MVC+DRV/r] and the [FTC/TDF+DRV/r] treatment arms, with two-sided 95% confidence interval, is shown for those patients who were R5 by genotype (including all who were originally randomized to ESTA and were R5 by genotype upon retesting), via the maximum likelihood (ML) method; Test type: Superiority or Other; Treatment difference = -0.0750, 95% CI 2-sided [-0.1343 to -0.0157], Standard Error of Mean 0.0303

10. Secondary Outcome: Virologic Outcomes at Week 48 Using Protocol-Defined Treatment Failure (PDTF).
Description: Per the protocol participants who meet the following criteria were regarded as PDTFs requiring a confirmatory plasma HIV-1 RNA determination: • Decrease in plasma HIV-1 RNA <1 log10 from baseline after Week 4 unless plasma HIV-1 RNA is <50 copies/mL, or • Plasma HIV-1 RNA >1.0 log10 above the nadir value after Week 4 where the nadir is the lowest plasma HIV-1 RNA concentration, or • Plasma HIV-1 RNA ≥50 copies/mL at any time after Week 24, or • Plasma HIV-1 RNA ≥50 copies/mL after suppression to <50 copies/mL on two consecutive visits, or • Decrease in plasma HIV-1 RNA ≤2 log10 from baseline on or after Week 12 unless plasma HIV-1 RNA is <400 copies/mL. Decrease in plasma HIV-1 RNA ≤2 log10 from baseline on or after Week 12 unless plasma HIV-1 RNA is <50 copies/mL (before August 30 2012) or <400 copies/mL (after August 30 2012).
Time Frame: Week 48
Population: The FAS consisted of all randomized participants who received at least one dose of the study drug. No imputation for missing values was performed for this endpoint. 'Evaluability' is determined by the on-treatment viral load (≥400 copies/mL at sample time point).
Measure: Number; unit: Number of participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
Number of participants
  Confirmed PDTF | 40 | 13
  Evaluable PDTF | 17 | 3

11. Secondary Outcome: Tropism Change Between Screening or Baseline and PDTF
Description: For participants meeting the PDTF criteria, tropism was assessed using the original randomized and alternate assays (ie, both genotype testing and ESTA). Data reported here corresponds to the timepoint at or after PDTF.
Time Frame: Week 48
Population: Number of Evaluable PDTF = Virology Analysis Population (VAP) 'Evaluability' is determined by the on-treatment viral load (≥400 copies/mL at sample time point).
Measure: Number; unit: participants
Groups:
- MVC+DRV/r - Baseline: Participants infected with R5 HIV-1 received oral tablets of Maraviroc 150 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for emtricitabine/tenofovir once daily. Summary of tropism results by baseline.
- MVC+DRV/r - Failure: Participants infected with R5 HIV-1 received oral tablets of Maraviroc 150 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for emtricitabine/tenofovir once daily. Summary of tropism results corresponding to timepoint at or after PDTF.
- FTC/TDF+DRV/r - Baseline: Participants infected with R5 HIV-1 received oral tablets of emtricitabine/tenofovir 200/300 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for maraviroc once daily. Summary of tropism results by baseline.
- FTC/TDF+DRV/r - Failure: Participants infected with R5 HIV-1 received oral tablets of emtricitabine/tenofovir 200/300 mg once daily plus darunavir/ritonavir 800/100 mg once daily plus placebo for maraviroc once daily. Summary of tropism results corresponding to timepoint at or after PDTF.
Arm/Group | MVC+DRV/r - Baseline | MVC+DRV/r - Failure | FTC/TDF+DRV/r - Baseline | FTC/TDF+DRV/r - Failure
Number analyzed (Participants) | 17 | 17 | 3 | 3
participants
  R5 (Randomized Assay) | 14 | 13 | 2 | 1
  NON R5 (Randomized Assay) | 1 | 1 | 0 | 0
  NR (Randomized Assay) | 2 | 3 | 1 | 2
  R5 (Alternate Assay) | 10 | 10 | 3 | 2
  NON R5 (Alternate Assay) | 2 | 3 | 0 | 1
  NR (Alternate Assay) | 5 | 4 | 0 | 0

12. Secondary Outcome: Number of Participants With Viral Resistance to Maraviroc (Maraviroc Treated Participants Only) in Participants Meeting PDTF Criteria.
Description: For participants meeting the PDTF criteria, viral resistance to maraviroc for maraviroc treated participants was assessed in patients with R5 virus at failure. The resistance level is calculated by reference to a laboratory strain of virus that is analyzed in parallel with the clinical isolate to identify 50% inhibitory concentrations (IC50). The maximal percent inhibition is the percent inhibition that is achieved in a titration of the drug at high concentrations when the addition of more drug does not result in increased inhibition. Maximal percent inhibition is obtained in the same way as the titration for IC50, but the key measure is of the plateau height of percent inhibition, where increased concentration of maraviroc does not result in additional inhibition. This is consistent with the virus developing some ability to use maraviroc-bound CCR5 for entry. A significant change in IC50 is not required for this mechanism.
Time Frame: Week 48
Population: The FAS consisted of all randomized participants who received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 17 | 3
participants
  Not eligible for analysis (failed tropism test) | 4 | 1
  Not eligible for analysis (non-R5 tropism) | 1 | 1
  Eligible for analysis (R5 virus using ESTA) | 12 | 1
  Results reported | 12 | 1
  Maximal percent inhibition <95% | 0 | 0
  IC50 FC ≥3.0 | 0 | 0

13. Secondary Outcome: Number of Participants With Resistance to Nucleoside/Nucleotide Reverse Transcriptase Inhibitors (NRTI), Non-nucleoside Reverse Transcriptase Inhibitors (NNRTI), and Protease Inhibitors (PI) in Participants Meeting PDTF Criteria
Description: For participants meeting the PDTF criteria, viral resistance (both genotypic and phenotypic) to NRTI, NNRTI, and PI's were assessed at Baseline and on-treatment. The assessment was performed using the overall (i.e. net) susceptibility score provided using the PhenoSense GT assay. The number of participants with successful assessments were 15/17 for the MVC+DRV/r arm and 3/3 for the FTC/TDF+DRV/r arm.
Time Frame: Week 48
Population: The FAS consisted of all randomized participants who received at least one dose of the study drug. The assessment was performed using the overall (ie. net) susceptibility score provided using the PhenoSense GT assay. The number of participants with successful assessments were 15 for the MVC+DRV/r arm and 3 for the FTC/TDF+DRV/r arm.
Measure: Number; unit: participants
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 15 | 3
participants
  NRTI - All (Baseline, n=15, 3) | 0 | 0
  NNRTI Delavirdine (Baseline, n=15, 3) | 1 | 0
  NNRTI Nevirapine (Baseline, n=15, 3) | 1 | 0
  NNRTI Efavirenz (Baseline, n=15, 3) | 1 | 0
  PRI - All (Baseline, n=15, 3) | 0 | 0
  NRTI - All (PDTF, n=15, 3) | 0 | 0
  NNRTI Delavirdine (PDTF, n=15, 3) | 1 | 0
  NNRTI Nevirapine (PDTF, n=15, 3) | 1 | 0
  NNRTI Efavirenz (PDTF, n=15, 3) | 1 | 0
  PRI - All (PDTF, n=15, 3) | 0 | 0

14. Secondary Outcome: Absolute Change From Baseline in Immune Cell Function at Week 48: Lymphocyte Marker Cluster of Differentiation 4 (CD4, Cell/mm^3)
Description: The differences in the magnitude of changes in CD4+ at Baseline and at Week 48 for maraviroc versus emtricitabine/tenofovir were compared.
Time Frame: Baseline, Week 48
Population: The FAS consisted of all randomized participants who received at least one dose of the study drug. Missing values were imputed using LOCF approach. Baseline was calculated as the average of all the pre-dose measurements excluding the screening value. If all pre-dose values were missing, screening value was considered as the baseline.
Measure: Mean (Standard Deviation); unit: cell/mm^3
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
cell/mm^3
  Baseline (n=396, 401) | 382.0 (173.4) | 379.5 (170.9)
  Week 48 (n=394, 396) | 576.9 (226.0) | 574.6 (232.1)
  Change from Baseline at Week 48 (n=394, 396) | 194.9 (175.5) | 194.2 (175.8)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; Results were from an ANCOVA model with change from Baseline as the response variable and the following fixed effect model terms: Treatment group, Screening plasma HIV RNA concentration, Screening Tropism Assay, Baseline value of the response variable; Test type: Superiority or Other; p = 0.9750, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-24.4 to 23.6]

15. Secondary Outcome: Percent Change From Baseline in Immune Cell Function at Week 48: Lymphocyte Activation Marker CD4 (%)
Description: The differences in the magnitude of changes in CD4+ from Baseline through Week 48 for maraviroc versus emtricitabine/tenofovir were compared.
Time Frame: Baseline, Week 48
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
Percentage of lymphocytes
  Baseline (n=396, 401) | 24.2 (7.9) | 24.5 (8.2)
  Week 48 (n=394, 396) | 31.3 (8.3) | 33.7 (8.6)
  Change from Baseline at Week 48 (n=394, 396) | 7.0 (5.7) | 9.2 (6.0)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; Results were from ANCOVA model with change from Baseline as the response variable and the following fixed effect model terms: Treatment group, Screening plasma HIV RNA concentration, Screening Tropism Assay, Baseline value of the response variable; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.1 to -1.5]

16. Secondary Outcome: Absolute Change From Baseline in Immune Cell Function at Week 48: Lymphocyte Marker Cluster of Differentiation 8 (CD8, Cell/mm^3)
Description: The differences in the magnitude of changes in CD8+ cell counts from baseline through Week 48 for maraviroc versus emtricitabine/tenofovir were compared.
Time Frame: Baseline, Week 48
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: cell/mm^3
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
cell/mm^3
  Baseline (n=396, 401) | 954.4 (502.1) | 914.5 (473.0)
  Week 48 (n=394, 396) | 900.0 (508.3) | 751.1 (386.7)
  Change from Baseline at Week 48 (n=394, 396) | -49.9 (410.7) | -157.9 (444.0)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 127.7, 95% CI 2-sided [76.5 to 178.8]

17. Secondary Outcome: Percent Change From Baseline in Immune Cell Function at Week 48: Lymphocyte Activation Marker CD8 (%)
Description: as for outcome 16
Time Frame: Baseline, Week 48
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
Percentage of lymphocytes
  Baseline (n=396, 401) | 57.0 (10.7) | 55.8 (10.5)
  Week 48 (n=394, 396) | 46.0 (10.4) | 43.0 (10.2)
  Change from Baseline at Week 48 (n=394, 396) | -10.9 (7.2) | -12.6 (8.1)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [1.1 to 3.1]

18. Secondary Outcome: Absolute Change in CD4+/CD8+ Ratio From Baseline to Week 48
Description: The differences in the magnitude of changes in CD4+/CD8+ ratio from Baseline through Weeks 48 for maraviroc versus emtricitabine/tenofovir were compared.
Time Frame: Baseline, Week 48
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 396 | 401
Ratio
  Baseline (n=396, 401) | 0.47 (0.24) | 0.48 (0.25)
  Week 48 (n=394, 396) | 0.75 (0.34) | 0.87 (0.45)
  Change from Baseline at Week 48 (n=394, 396) | 0.28 (0.22) | 0.39 (0.34)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; Results are from an ANCOVA model with change from Baseline as the response variable and the following fixed effect model terms: Treatment group, Screening plasma HIV RNA concentration, Screening Tropism Assay, Baseline value of the response variable; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.15 to -0.07]

19. Secondary Outcome: Changes in Peripheral Fat Distribution Using Dual Energy X-ray Absorptiometry [DEXA] Scan From Baseline and at Week 48.
Description: A sub-study was conducted in which the participants underwent whole-body DEXA scans to evaluate peripheral fat tissue estimates for left and right arms and legs and truncal fat mass and truncal lean mass. Truncal abdominal fat were estimated from the DEXA scan field set on the torso. The effects on estimates of fat mass and lean mass were addressed by providing LSMs of change from baseline.
Time Frame: Week 48
Population: Safety Analysis Set was the same as the FAS consisting of all randomized participants who received at least one dose of the study drug but analyzed as realized for tropism assay and treatment. Missing values were imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: gram
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 52 | 56
gram | -181.6 (569.8) | -257.5 (556.9)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; Results are from ANCOVA model with change from Baseline as the response variable and the following fixed effect model terms: treatment group, age, race, Screening BMI, and Baseline value of the response variable. Treatment differences are estimated using LS means with factor levels weighted according to overall analysis population proportions; Test type: Superiority or Other; p = 0.8379, ANCOVA; Mean Difference (Final Values) = 75.861, 95% CI 2-sided [-658.181 to 809.903]

20. Secondary Outcome: Changes in Trunk to Limb Fat Distribution Using DEXA Scan From Baseline and at Week 48
Description: as for outcome 19
Time Frame: Week 48
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 52 | 56
ratio | 0.017 (0.048) | -0.014 (0.048)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.3376, ANCOVA; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.033 to 0.094]

21. Secondary Outcome: Changes in Bone Mineral Density (Using DEXA Scan and Serum Markers) From Baseline and at Week 48 - Total Hip BMD
Description: Bone mineral density was evaluated by DEXA scan in a subset of participants who consented to these evaluations. The effects on BMD were addressed by providing LSMs of change from baseline bone mineral density of the lumbar spine (L1-L4), left total hip and femoral neck as measured by the DEXA scan.
Time Frame: Week 48
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 47 | 57
g/cm^2 | -0.014 (0.005) | -0.028 (0.005)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.0043, ANCOVA; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [0.004 to 0.023]

22. Secondary Outcome: Changes in Bone Mineral Density (Using DEXA Scan and Serum Markers) From Baseline and at Week 48 - Femoral Neck BMD
Description: Bone mineral density was evaluated by DEXA scan in a subset of participants who consented to these evaluations. The effects on BMD were addressed by providing LSMs of change from Baseline bone mineral density femoral neck as measured by the DEXA scan.
Time Frame: Week 48
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 47 | 57
g/cm^2 | -0.021 (0.007) | -0.029 (0.007)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.2273, ANCOVA; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.005 to 0.022]

23. Secondary Outcome: Changes in Bone Mineral Density (Using DEXA Scan and Serum Markers) From Baseline and at Week 48 - AP Lumbar Spine (L1 - L4) BMD
Description: Bone mineral density was evaluated by DEXA scan in a subset of participants who consented to these evaluations. The effects on BMD were addressed by providing LSMs of change from baseline bone mineral density of the lumbar spine (L1-L4) as measured by the DEXA scan.
Time Frame: Week 48
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 54 | 60
g/cm^2 | -0.020 (0.006) | -0.025 (0.006)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.4188, ANCOVA; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.007 to 0.018]

24. Secondary Outcome: Change in Bone Turnover Markers From Baseline and at Week 48 - Blood Osteocalcin
Description: Bone turnover marker, osteocalcin, was collected in the subset of participants participating in the DEXA scan sub-study.
Time Frame: Week 48
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 52 | 61
ng/mL | 5.61 (8.02) | 6.77 (8.31)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.1722, ANCOVA; Mean Difference (Final Values) = -2.12, 95% CI 2-sided [-5.17 to 0.94]

25. Secondary Outcome: Change in Bone Turnover Markers From Baseline and at Week 48 - Type 1 Collagen Peptide (CTX-1)
Description: Bone turnover marker, C-telopeptide of type 1 collagen (CTx), was collected in the subset of participants participating in the DEXA scan sub-study.
Time Frame: Week 48
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Number analyzed (Participants) | 53 | 62
pg/mL | 121.13 (243.03) | 223.52 (293.03)
Statistical Analysis 1: Comparison: MVC+DRV/r vs FTC/TDF+DRV/r; Results are from an ANCOVA model with change from Baseline as the response variable and the following fixed effect model terms: treatment group, age, race, Screening BMI, Baseline value of the response variable. Treatment differences are estimated using LS means with factor levels weighted according to overall analysis population proportions; Test type: Superiority or Other; p = 0.0071, ANCOVA; Mean Difference (Final Values) = -126.78, 95% CI 2-sided [-218.34 to -35.23]

ADVERSE EVENTS:
Time Frame: From the day the first dose of the study drug was administered to 28 days after the last dose of the study drug was administered.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | MVC+DRV/r | FTC/TDF+DRV/r
Serious Adverse Events (participants affected / at risk) | 41/396 | 40/401
Other Adverse Events (participants affected / at risk) | 257/396 | 285/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MVC+DRV/r (N=396) | FTC/TDF+DRV/r (N=401)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 1
Hernia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Acute hepatitis C (Infections and infestations) | 0 | 2
Anal abscess (Infections and infestations) | 1 | 1
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Eye infection syphilitic (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 1
Lymph node abscess (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 2
Amylase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Drug dependence (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Drug rehabilitation (Surgical and medical procedures) | 0 | 2
Papilloma excision (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Shigella infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 2
Mental disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anal lesion excision (Surgical and medical procedures) | 0 | 1
THROMBUS, AORTIC HEPATIC ARTERY (Hepatobiliary disorders) | 0 | 1 — BEING QUERIED
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Herpes zoster infection neurological (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MVC+DRV/r (N=396) | FTC/TDF+DRV/r (N=401)
Diarrhoea (Gastrointestinal disorders) | 88 | 135
Nausea (Gastrointestinal disorders) | 34 | 45
Fatigue (General disorders) | 27 | 46
Bronchitis (Infections and infestations) | 25 | 24
Gastroenteritis (Infections and infestations) | 23 | 16
Nasopharyngitis (Infections and infestations) | 48 | 55
Upper respiratory tract infection (Infections and infestations) | 40 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 23
Headache (Nervous system disorders) | 27 | 47
Depression (Psychiatric disorders) | 26 | 29
Insomnia (Psychiatric disorders) | 15 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 30
Rash (Skin and subcutaneous tissue disorders) | 37 | 30
Abdominal distension (Gastrointestinal disorders) | 9 | 22
Influenza (Infections and infestations) | 22 | 20
Syphilis (Infections and infestations) | 15 | 23
Blood cholesterol increased (Investigations) | 22 | 10
Low density lipoprotein increased (Investigations) | 22 | 11

LIMITATIONS AND CAVEATS:
The study was terminated following a preliminary review of the 48- week primary clinical efficacy data by the study's external independent Data Monitoring Committee's recommendation based on inferior efficacy of the investigational MVC+DRV/r arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.